CLINICAL TRIAL: NCT04637451
Title: The Comparison of the Efficacy of Gingival Unit Graft With Connective Tissue Graft in Root Coverage: A Randomized Split-Mouth Clinical Trial
Brief Title: The Comparison of the Efficacy of Gingival Unit Graft With Connective Tissue Graft in Root Coverage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Sibel Kayaalti-Yuksek, Assistant Professor, Okan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/174
Record Dates: First submitted 2020-11-10; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Gingival Recession; Periodontal Diseases
MeSH Terms: conditions — Gingival Recession; Periodontal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gingival Unit Graft (Experimental): For test group, gingival recessions were treated with gingival unit graft.
  Interventions: Procedure: Root coverage treatment
- Connective Tissue Graft (Other): For Control group, gingival recessions were treated with connective tissue graft.
  Interventions: Procedure: Root coverage treatment

INTERVENTIONS:
Procedure: Root coverage treatment — Gingival unit graft Connective tissue graft

SUMMARY:
The purpose of the study is to compare the clinical effectiveness of gingival unit graft (GUG) and connective tissues graft (CTG) in Miller's class I and II gingival recession.

DETAILED DESCRIPTION:
Patients who accept the study have provided information about the study and required a written informed consent form. The clinical effectiveness of two different periodontal surgical techniques (gingival unit graft and connective tissue graft) in gingival recessions will be evaluated. Periodontal measurements (gingival recession, keratinized gingiva height) and patient-reported outcomes (intra and post-operative pain, patient satisfaction and hypersensitivity) are defined.

ELIGIBILITY:
Inclusion Criteria:

* Systemic healthy individuals
* Presence Miller's class I and II gingival recession in the anterior and premolar teeth

Exclusion Criteria:

* Age <18 years
* Pregnancy
* Lactation
* Any cardiovascular, renal or hepatic conditions
* History of periodontal surgery
* Tooth mobility
* Presence of probing depth >3 mm and caries or restorations in the teeth undergoing treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-07-15 (Actual); Study Completion 2016-07-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Gingival Recession Depth at 6 month | Baseline and month 6.
  The gingival recession depth consists of the distance from the cement-enamel junction to the most apical extension of the gingival margin. The measurement is recorded in millimeters. Change= (6 month score-baseline score)
Change from Baseline Keratinized Gingiva Height at 6 month | Baseline and month 6.
  Keratinized gingiva height, measured as the distance from the gingival margin to the mucogingival line. The measurement is recorded in millimeters. Change= (6 month score-baseline score)

SECONDARY OUTCOMES:
Change from Baseline Root Hypersensitivity at 6 month | Baseline and month 6.
  Root hypersensitivity at baseline and post-operative 6 month utilizing a visual numerical scale (VNS) test are defined. Possible scores range from (0=no sensitive and 10= worst possible sensitive). Change= (6 month score-baseline score)
Change from Baseline Patient Satisfaction at 6 month | Baseline and month 6.
  The patient satisfaction with the gingiva position, structure and color of the gingival recessions sites utilizing a VNS test (0=not satisfied and 10=very satisfied) are defined. Possible scores range from 0 (not satisfied) to 10 (very satisfied). Change= (6 month score-baseline score)
Change from Baseline Pain at 1 week | Baseline and week 1.
  Pain perception of the surgery at intra and post-operative period (week 1) utilizing a VNS test are defined. Possible scores range from 0 (no pain) to 10 (worst possible pain). Change= (1 week score-baseline score)
Change from Baseline Pain at 2 week | Baseline and week 2.
  Pain perception of the surgery at intra and post-operative period (week 2) utilizing a VNS test are defined. Possible scores range from 0 (no pain) to 10 (worst possible pain). Change= (2 week score-baseline score)

CONTACTS AND LOCATIONS:
Locations (1):
- Sibel Kayaaltı Yüksek, Istanbul, Tuzla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zucchelli G, Mounssif I. Periodontal plastic surgery. Periodontol 2000. 2015 Jun;68(1):333-68. doi: 10.1111/prd.12059. PMID 25867992
- [Background] Cairo F, Pagliaro U, Buti J, Baccini M, Graziani F, Tonelli P, Pagavino G, Tonetti MS. Root coverage procedures improve patient aesthetics. A systematic review and Bayesian network meta-analysis. J Clin Periodontol. 2016 Nov;43(11):965-975. doi: 10.1111/jcpe.12603. Epub 2016 Sep 16. PMID 27454460
- [Background] Allen AL. Use of the gingival unit transfer in soft tissue grafting: report of three cases. Int J Periodontics Restorative Dent. 2004 Apr;24(2):165-75. PMID 15119887
- [Background] Kuru B, Yildirim S. Treatment of localized gingival recessions using gingival unit grafts: a randomized controlled clinical trial. J Periodontol. 2013 Jan;84(1):41-50. doi: 10.1902/jop.2012.110685. Epub 2012 Mar 5. PMID 22390550
- [Background] Yildirim S, Kuru B. Gingival unit transfer using in the Miller III recession defect treatment. World J Clin Cases. 2015 Feb 16;3(2):199-203. doi: 10.12998/wjcc.v3.i2.199. PMID 25685769
- [Background] Del Pizzo M, Modica F, Bethaz N, Priotto P, Romagnoli R. The connective tissue graft: a comparative clinical evaluation of wound healing at the palatal donor site. A preliminary study. J Clin Periodontol. 2002 Sep;29(9):848-54. doi: 10.1034/j.1600-051x.2002.290910.x. PMID 12423299
- [Background] Douglas de Oliveira DW, Oliveira-Ferreira F, Flecha OD, Goncalves PF. Is surgical root coverage effective for the treatment of cervical dentin hypersensitivity? A systematic review. J Periodontol. 2013 Mar;84(3):295-306. doi: 10.1902/jop.2012.120143. Epub 2012 May 1. PMID 22548583
- [Background] Camargo PM, Melnick PR, Kenney EB. The use of free gingival grafts for aesthetic purposes. Periodontol 2000. 2001;27:72-96. doi: 10.1034/j.1600-0757.2001.027001072.x. No abstract available. PMID 11551301
- [Derived] Kayaalti-Yuksek S, Yaprak E. The comparison of the efficacy of gingival unit graft with connective tissue graft in recession defect coverage: a randomized split-mouth clinical trial. Clin Oral Investig. 2022 Mar;26(3):2761-2770. doi: 10.1007/s00784-021-04252-5. Epub 2021 Nov 17. PMID 34787718